CLINICAL TRIAL: NCT03849430
Title: Longitudinal Analysis of the Health-related Quality of Life in Glioma Patients and Setting Up a Large-scale, Prospective Database for Glioma Patients Treated in UZ Leuven
Brief Title: Longitudinal Analysis of the Health-related Quality of Life in Glioma Patients
Acronym: Glioma2015
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof. Dr. Steven De Vleeschouwer, Member of Staff Neurosurgery, Clinical Professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S58343
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Glioma of Brain
Keywords: Low grade glioma; High grade glioma; HRQOL
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Gliomas are the most common primary intracranial tumors, representing at least 75% of all primary malignant brain tumors. Histopathologically, gliomas are classified into different subgroups including astrocytomas (60-70%), oligodendrogliomas (10-30%), ependymomas (<10%) and mixed gliomas (i.e. oligoastrocytomas) depending on the cell type from which they originate. The World Health Organization currently classifies gliomas based on histopathological analysis in which the presence (or absence) and the degree of specific histopathological features determines the grade of malignancy. Grade I (pilocytic astrocytoma) and grade II (diffuse astrocytoma, oligodendroglioma, mixed oligoastrocytoma, and pleomorphic xanthoastrocytoma) are termed low-grade gliomas (LGGs), whereas grade III (anaplastic astrocytoma, anaplastic oligodendroglioma or anaplastic oligoastrocytoma) and grade IV (glioblastoma) represent high-grade gliomas (HGGs).

Given the incurable nature of gliomas, the maintenance or improvement of the patient's quality of life are extremely important. The benefits of multimodal treatment strategies, in terms of prolonged survival or delay of progression, have to be carefully balanced against the side effects of the treatment, which may adversely influence patient's functioning and well-being during his/her remaining life span.

Measuring a brain tumor patients functioning and well-being goes far beyond assessing (progression-free) survival or tumor response to treatment on imaging. A more integrated way to measure patients functioning and well-being is the assessment of a patient's health-related quality of life (HRQOL). HRQOL is defined as a personal self-assessed ability to function in the physical, psychological, emotional, and social domains of day-to-day life.

The main goal of this study is to perform a large-scale, prospective and long-term analysis of the HRQOL in patients diagnosed with glioma.

DETAILED DESCRIPTION:
Aims of the study

The main goal of this study is to perform a large-scale, prospective and long-term analysis of the HRQOL in patients diagnosed with glioma and to set up a database which contains general patient characteristics, tumor information, treatment strategy and follow-up data of each included patient. This large-scale database will allow the investigator to investigate several relevant research questions in a well-documented group of glioma patients.

Methodology

HRQOL is a multidimensional concept covering physical, psychological and social domains as well as symptoms induced by the disease and the treatment. Currently there is no single gold standard tool to measure HRQOL, and several valid measures of HRQOL in brain tumor patients are available. In this study the investigator will use the EQ-5D questionnaire to report patient's HRQOL. The EQ-5D is widely used and has been validated in many different patient populations. It has been designed so that patients can describe the extent to which they have a problem in each of the five dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression The timing of the HRQOL questionnaires will depend on whether a patient will be diagnosed with either a LGG or a HGG. Moreover, as the current treatment strategies for LGG patients and for relapsed HGG patients are highly variable, the investigator scheduled the HRQOL measurements not in function of the treatment, but rather in function of the classical, standard-of-care patient follow-up (either 3 or 6 monthly).

Missing data

When there are missing data for some patients, the question arises as to whether patients with missing data differ from those who returned completed forms. As a consequence, missing data presents problems in the analysis and the interpretation of the results. Hence, the amount of missing data should be minimized. A regular check on missing data will be performed by the CTA. In case the HRQOL form was not completed by the included patient, the patient will be contacted by phone or e-mail and he/she will be asked to provide an answer to the different questions of the HRQOL questionnaire in order to avoid missing data. In case the patient is unable to complete the HRQOL questionnaire, the CTA will report the reason for non-completion in the database.

ELIGIBILITY:
Inclusion criteria:

* age ≥ 18 years
* patients diagnosed and treated for a high- or low grade glioma
* treatment in UZ Leuven

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The GLIOMA-2015 study will include adult patients that will be diagnosed and/or operated and/or treated and followed-up for a low- or high grade glioma in UZ Leuven.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2015-12-14 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Change over time of quality of life from diagnosis until end of active treatment | Every 3 months, from diagnosis until date of decease or up to 10 year, whichever came first
  Quality of life is assessed using the EQ-5D-5L (EuroQol 5 Dimensions 5 Level scale), which has 2 components. The description component measures health status in terms of 5 dimensions; mobility (ability to walk), self-care (ability to wash or dress by oneself), usual activities (performance in work, study, housework, family or leisure activities), pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The respondents self-rate their level of severity for each dimension. Each level of each dimension corresponds to a 1-digit number. All together a 5-digit number describes the patient's health state (3,125 (55) different health states are possible). In the evaluation component, the respondents evaluate their overall health status by valuing health-related quality of life from 0 (corresponding to the worst health you can imagine) to 100 (corresponding to the best health you can imagine).
Survival | At time of decease or up to 10 year
  Date of decease will be reported in a prospective database

SECONDARY OUTCOMES:
Treatment strategy | From date of first diagnoses until date of decease or up to 10 year, whichever came first
  All treatment details will be reported in a prospective database

CONTACTS AND LOCATIONS:
Overall Officials: Steven De Vleeschouwer, MD Phd, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No